CLINICAL TRIAL: NCT04291560
Title: Promoting Stretching Exercise to Reduce Cardiovascular Health Risk in Late Pregnant Women With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18-3091; 1R01NR017944-01A1 (NIH)
Record Dates: First submitted 2020-02-21; First posted 2020-03-02 (Actual); Results first posted 2025-11-17 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-01

CONDITIONS: Pregnancy Related; Cardiovascular Risk Factor; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: A parallel design will be used, with an equal allocation of 306 obese pregnant women to the two groups: stretching exercise and enhanced usual care.
Who Masked: Outcomes Assessor
Masking Description: Masking will not be completed in this trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prenatal Heart Smart Intervention (Experimental): This group will have usual care completed and supportive calls from a facilitator to discuss adherence to the home exercise. In addition, the group will complete a sequential static stretching exercise 5 days per week for 10 weeks. The stretching exercise consists of 20 seconds of stretching, for 3 repetitions per muscle group.
  Interventions: Behavioral: Stretching Exercise Intervention
- Usual Care (Control) (No Intervention): This group will have usual care completed and supportive calls from a facilitator to discuss adherence to the home exercise. In addition, this group will complete moderate-intensity walking 5 days per week for 10 weeks in accordance to usual care.

INTERVENTIONS:
Behavioral: Stretching Exercise Intervention — Sequential static stretching of the large skeletal muscle group 5 days per week. Each skeletal group is stretched for 20 seconds for 3 repetitions.
  Arms: Prenatal Heart Smart Intervention

SUMMARY:
The purpose of this trial is to determine whether a stretching intervention is superior to a usual care control condition (moderate/vigorous activity 30 minutes daily, 5 days per week) for pregnant women from 27 to 37 gestational weeks.

DETAILED DESCRIPTION:
Although being sedentary can lead to excess risk for maternal and child mortality and morbidity, most pregnant women reduce their physical activity and only 8% meet the recommendations in the 3rd trimester.

In a prior randomized control trial, it was found that fewer women who stretched developed preeclampsia than did women who walked (3/60 "stretchers" vs. 10/64 "walkers", p=.05).

In this study, participants will either receive a stretching intervention

ELIGIBILITY:
Inclusion Criteria:

* Pregnant at less than 24 weeks gestation
* Singleton pregnancy
* BMI ≥ 30 kg/m^2 at their first prenatal care visit
* English or Spanish speaking

Exclusion Criteria:

* Women who expect or are scheduled to deliver prior to 37 weeks gestation
* Women who expect to move from the area during their participation in the study
* Women who are unable to exercise for 30 or more minutes 3 times per week

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SeonAe Yeo, PhD, FAAN, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 224 participants consented during early pregnancy. After consenting, participants underwent a run-in period until reaching approximately 27 weeks gestation, at which point a baseline visit was scheduled. 108 participants completed this baseline visit, and thus were randomized to one of the study arms.
Period: Overall Study
Arm/Group | Prenatal Heart Smart Intervention | Usual Care (Control)
Started | 53 | 55
Completed | 53 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prenatal Heart Smart Intervention | Usual Care (Control) | Total
Number analyzed (Participants) | 53 | 55 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (3.7) | 31.0 (5.7) | 31.9 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 55 | 108
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 6 | 17
  Not Hispanic or Latino | 41 | 44 | 85
  Unknown or Not Reported | 1 | 5 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 19 | 41
  White | 24 | 27 | 51
  More than one race | 2 | 5 | 7
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53 | 55 | 108

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure From Baseline (27 Gestational Weeks) to 32 Gestational Weeks
Description: Average systolic blood pressure measurement between two measurements, assessed at baseline (approximately 27 gestational weeks) and approximately 5 weeks after baseline (approximately 32 gestational weeks). Three total measurements will be taken, the first will be removed and the second two averaged.
Time Frame: Baseline (approximately 27 gestational weeks) to approximately 5 weeks after baseline (approximately 32 gestational weeks)
Population: Only includes participants who completed blood pressure measures at their 32 week follow-up visit.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Prenatal Heart Smart Intervention | Usual Care (Control)
Number analyzed (Participants) | 33 | 39
mmHg | 0.73 (8.21) | -1.56 (8.34)

2. Primary Outcome: Change in Systolic Blood Pressure From Baseline (27 Gestational Weeks) to 37 Gestational Weeks
Description: Average systolic blood pressure measurement between two measurements, assessed at baseline (approximately 27 gestational weeks) and approximately 10 weeks after baseline (approximately 37 gestational weeks). Three total measurements will be taken, the first will be removed and the second two averaged.
Time Frame: Baseline (approximately 27 gestational weeks) to approximately 10 weeks after baseline (approximately 37 gestational weeks)
Population: Only includes participants who completed blood pressure measures at their 37 week follow-up visit.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Prenatal Heart Smart Intervention | Usual Care (Control)
Number analyzed (Participants) | 28 | 28
mmHg | 3.14 (8.02) | 6.23 (10.07)

3. Primary Outcome: Change in Diastolic Blood Pressure From Baseline (27 Gestational Weeks) to 32 Gestational Weeks
Description: Average diastolic blood pressure measurement between two measurements, assessed at baseline (approximately 27 gestational weeks) and approximately 5 weeks after baseline (approximately 32 gestational weeks) Three total measurements will be taken, the first will be removed and the second two averaged.
Time Frame: as for outcome 1
Population: Only includes participants who completed blood pressure measures at their 32 week follow-up visit.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Prenatal Heart Smart Intervention | Usual Care (Control)
Number analyzed (Participants) | 33 | 39
mmHg | 0.41 (7.75) | 1.42 (5.28)

4. Primary Outcome: Change in Diastolic Blood Pressure From Baseline (27 Gestational Weeks) to 37 Gestational Weeks
Description: Average diastolic blood pressure measurement between two measurements, assessed at baseline (approximately 27 gestational weeks) and approximately 10 weeks after baseline (approximately 32 gestational weeks). Three total measurements will be taken, the first will be removed and the second two averaged.
Time Frame: as for outcome 2
Population: Only includes participants who completed blood pressure measures at their 37 week follow-up visit.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Prenatal Heart Smart Intervention | Usual Care (Control)
Number analyzed (Participants) | 28 | 28
mmHg | 4.52 (7.08) | 7.63 (7.27)

5. Primary Outcome: Change in Sympatho-vagal Balance Projection Period (PEP) for Sympathetic Activity From Baseline (27 Gestational Weeks) to 32 Gestational Weeks
Description: The time in milliseconds from the ECG R point (left ventricular depolarization) and the B-point on the Dz/dt wave form (opening of the aortic valve), assessed at baseline (27 gestational weeks) and 32 gestational weeks.
Time Frame: as for outcome 1
Population: This variable required cardiac impedance data, which were not collected from any participants. PEP was initially proposed as a measure of autonomic function; however, we were already collecting high-frequency (HF) heart rate variability, a more well-established indicator of autonomic function. Adding another measure was deemed an unnecessary burden on participants, so it was removed from the protocol.
Arm/Group | Prenatal Heart Smart Intervention | Usual Care (Control)
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Change in Sympatho-vagal Balance Projection Period (PEP) for Sympathetic From Baseline (27 Gestational Weeks) to 37 Gestational Weeks
Description: The time in milliseconds from the ECG R point (left ventricular depolarization) and the B-point on the Dz/dt wave form (opening of the aortic valve), assessed at baseline (27 gestational weeks) and 37 gestational weeks.
Time Frame: as for outcome 2
Population: as for outcome 5
Arm/Group | Prenatal Heart Smart Intervention | Usual Care (Control)
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Change in High Frequency of Heart Rate Variability From Baseline (27 Gestational Weeks) to 32 Gestational Weeks
Description: High frequency of heart rate variability (log(ms^2/Hz)) from an electrocardiogram, assessed at baseline (27 gestational weeks) and 32 gestational weeks.
Time Frame: as for outcome 1
Population: Only includes participants who completed heart rate variability measures at their 32 week follow-up visit.
Measure: Mean (Standard Deviation); unit: log(ms^2/Hz)
Arm/Group | Prenatal Heart Smart Intervention | Usual Care (Control)
Number analyzed (Participants) | 30 | 41
log(ms^2/Hz) | -0.13 (1.42) | -0.03 (1.48)

8. Primary Outcome: Change in High Frequency of Heart Rate Variability From Baseline (27 Gestational Weeks) to 37 Gestational Weeks
Description: High frequency of heart rate variability (log(ms^2/Hz)) from an electrocardiogram, assessed at baseline (27 gestational weeks) and 37 gestational weeks.
Time Frame: as for outcome 2
Population: Only includes participants who completed heart rate variability measures at their 37 week follow-up visit.
Measure: Mean (Standard Deviation); unit: log(ms^2/Hz)
Arm/Group | Prenatal Heart Smart Intervention | Usual Care (Control)
Number analyzed (Participants) | 27 | 25
log(ms^2/Hz) | -0.42 (1.02) | -0.37 (1.27)

9. Primary Outcome: Change in Arterial Stiffness Assessed by SphygmoCor XCEL From Baseline (27 Gestational Weeks) to 32 Gestational Weeks
Description: Carotid-femoral pulse wave velocity (PWV) is a measure of arterial stiffness reported in m/s. Lower values reflect less arterial stiffness.
Time Frame: as for outcome 1
Population: Only includes participants who completed PWV measures at their 32 week follow-up visit.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Prenatal Heart Smart Intervention | Usual Care (Control)
Number analyzed (Participants) | 27 | 34
m/s | 0.20 (1.81) | 0.19 (0.78)

10. Primary Outcome: Change in Arterial Stiffness Assessed by SphygmoCor XCEL From Baseline (27 Gestational Weeks) to 37 Gestational Weeks
Description: as for outcome 9
Time Frame: as for outcome 2
Population: Only includes participants who completed PWV measures at their 37 week follow-up visit.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Prenatal Heart Smart Intervention | Usual Care (Control)
Number analyzed (Participants) | 24 | 22
m/s | 0.07 (1.34) | 0.59 (0.99)

11. Secondary Outcome: Onset of Preeclampsia Anytime Between Baseline (27 Weeks Gestation) and the End of Pregnancy
Description: Presence of preeclampsia anytime between baseline (27 weeks gestation) and the end of pregnancy in the electronic medical record.
Time Frame: Baseline (approximately 27 Weeks Gestation) to the End of Pregnancy (approximately 40 weeks); approximately 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal Heart Smart Intervention | Usual Care (Control)
Number analyzed (Participants) | 53 | 55
Participants | 4 | 7

12. Secondary Outcome: Onset of Eclampsia Anytime Between Baseline (27 Weeks Gestation) and the End of Pregnancy
Description: Presence of eclampsia anytime between baseline (27 weeks gestation) and the end of pregnancy in the electronic medical record.
Time Frame: Baseline (approximately 27 Weeks Gestation) to the End of Pregnancy (approximately 40 weeks); approximately 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal Heart Smart Intervention | Usual Care (Control)
Number analyzed (Participants) | 53 | 55
Participants | 0 | 0

13. Secondary Outcome: Onset of Pregnancy Induced Hypertension Anytime Between Baseline (27 Weeks Gestation) and the End of Pregnancy
Description: Presence of pregnancy induced hypertension anytime between baseline (27 weeks gestation) and the end of pregnancy in the electronic medical record.
Time Frame: Baseline (approximately 27 Weeks Gestation) to the End of Pregnancy (approximately 40 weeks); approximately 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal Heart Smart Intervention | Usual Care (Control)
Number analyzed (Participants) | 53 | 55
Participants | 15 | 21

14. Secondary Outcome: Onset of Gestational Diabetes Anytime Between Baseline (27 Weeks) and the End of Pregnancy
Description: Presence of gestational diabetes anytime between baseline (27 weeks gestation) and the end of pregnancy in the electronic medical record.
Time Frame: Baseline (approximately 27 Weeks Gestation) to the End of Pregnancy (approximately 40 weeks); approximately 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal Heart Smart Intervention | Usual Care (Control)
Number analyzed (Participants) | 53 | 55
Participants | 6 | 6

15. Secondary Outcome: Preterm Delivery at End of Pregnancy
Description: Presence of preterm delivery in the electronic medical record.
Time Frame: Baseline (approximately 27 Weeks Gestation) to the End of Pregnancy (approximately 40 weeks); approximately 13 weeks
Population: Only includes babies delivered within the hospital system to which the study team had record access, or where the mother provided basic delivery information to the study team post-delivery.
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal Heart Smart Intervention | Usual Care (Control)
Number analyzed (Participants) | 51 | 54
Participants | 3 | 2

16. Secondary Outcome: Elective or Emergency Cesarean Section at End of Pregnancy
Description: Presence of an elective or emergency cesarean section in the electronic medical record.
Time Frame: Baseline (approximately 27 Weeks Gestation) to the End of Pregnancy (approximately 40 weeks); approximately 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal Heart Smart Intervention | Usual Care (Control)
Number analyzed (Participants) | 53 | 55
Participants | 18 | 18

17. Secondary Outcome: Composite Score of Maternal Outcomes at the End of Pregnancy
Description: The composite score of maternal outcomes (onset of preeclampsia, eclampsia pregnancy induced hypertension, gestational diabetes, preterm delivery, and elective or emergency cesarean section) is obtained at the end of pregnancy. Scores range from 0-6, with higher scores indicating a less healthy pregnancy.
Time Frame: Baseline (approximately 27 Weeks Gestation) to the End of Pregnancy (approximately 40 weeks); approximately 13 weeks
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prenatal Heart Smart Intervention | Usual Care (Control)
Number analyzed (Participants) | 51 | 54
score on a scale | 0.90 (1.12) | 1.00 (1.05)

18. Secondary Outcome: Intrauterine Death at End of Pregnancy
Description: Presence of an intrauterine death in the electronic medical record.
Time Frame: Baseline (approximately 27 Weeks Gestation) to the End of Pregnancy (approximately 40 weeks); approximately 13 weeks
Population: Only includes babies delivered within the hospital system to which the study team had record access.
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal Heart Smart Intervention | Usual Care (Control)
Number analyzed (Participants) | 50 | 53
Participants | 0 | 0

19. Secondary Outcome: Child Being Small for Gestational Age at the End of Pregnancy
Description: Presence of the child being small for gestational age in the electronic medical record.
Time Frame: Baseline (approximately 27 Weeks Gestation) to the End of Pregnancy (approximately 40 weeks); approximately 13 weeks
Population: Only includes babies delivered within the hospital system to which the study team had record access.
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal Heart Smart Intervention | Usual Care (Control)
Number analyzed (Participants) | 50 | 53
Participants | 2 | 5

20. Secondary Outcome: Child Being Large for Gestational Age at the End of Pregnancy
Description: Presence of the child being large for gestational age in the electronic medical record.
Time Frame: Baseline (approximately 27 Weeks Gestation) to the End of Pregnancy (approximately 40 weeks); approximately 13 weeks
Population: Only includes babies delivered within the hospital system to which the study team had record access.
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal Heart Smart Intervention | Usual Care (Control)
Number analyzed (Participants) | 50 | 53
Participants | 7 | 11

21. Secondary Outcome: Neonatal Intensive Care Unit Admission at the End of Pregnancy
Description: Presence of a neonatal intensive care unit admission in the electronic medical record.
Time Frame: Baseline (approximately 27 Weeks Gestation) to the End of Pregnancy (approximately 40 weeks); approximately 13 weeks
Population: Only includes babies delivered within the hospital system to which the study team had record access.
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatal Heart Smart Intervention | Usual Care (Control)
Number analyzed (Participants) | 50 | 53
Participants | 1 | 1

22. Secondary Outcome: Composite Score of Fetal/Neonatal Outcomes at the End of Pregnancy.
Description: The composite score of fetal/neonatal outcomes (intrauterine death, child being small, child being large, neonatal intensive care admission) is obtained at the end of pregnancy. Scores range from 0-4, with higher scores indicating a less healthy fetus/neonate.
Time Frame: Baseline (approximately 27 Weeks Gestation) to the End of Pregnancy (approximately 40 weeks); approximately 13 weeks
Population: Only includes babies delivered within the hospital system to which the study team had record access.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prenatal Heart Smart Intervention | Usual Care (Control)
Number analyzed (Participants) | 50 | 53
score on a scale | 0.20 (0.40) | 0.32 (0.47)

ADVERSE EVENTS:
Time Frame: From the time of randomization (about 27 weeks gestation) through 8 weeks after delivery, an approximate total of 21 weeks.
Arm/Group | Prenatal Heart Smart Intervention | Usual Care (Control)
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/55
Serious Adverse Events (participants affected / at risk) | 5/53 | 8/55
Other Adverse Events (participants affected / at risk) | 35/53 | 41/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prenatal Heart Smart Intervention (N=53) | Usual Care (Control) (N=55)
Preeclampsia (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 7 (7)
Hospitalization for Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Fetal abnormality (abdominal mass) detected via ultrasound (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prenatal Heart Smart Intervention (N=53) | Usual Care (Control) (N=55)
Shortness of breath while exercising (Cardiac disorders) | 3 (3) | 3 (6)
Dizziness while exercising (Cardiac disorders) | 6 (6) | 2 (2)
Reported contracting respiratory virus (cold, flu, RSV, or Covid) (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 3 (3)
Gastrointestinal virus (Gastrointestinal disorders) | 3 (3) | 1 (1)
Pregnancy-related pain or soreness (Pregnancy, puerperium and perinatal conditions) | 6 (7) | 6 (6) — Includes hip pain, sciatica, back pain, abdominal soreness
Delivery via Caesarean section (Pregnancy, puerperium and perinatal conditions) | 18 (18) | 18 (18)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 15 (15) | 21 (21)
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 6 (6) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Original version (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT04291560/Prot_SAP_001.pdf
  • Study Protocol and Statistical Analysis Plan: Revised version to remove Cardiac Impedance measures (2025-10-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT04291560/Prot_SAP_002.pdf
  • Informed Consent Form (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/60/NCT04291560/ICF_000.pdf